CLINICAL TRIAL: NCT04837144
Title: Evaluation of the Safety and Usability of the MAK Exoskeleton in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MarsiBionics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAKStrokeUSII
Record Dates: First submitted 2020-11-03; First posted 2021-04-08 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Stroke; Gait, Hemiplegic
Keywords: exoskeleton; robotic device; gait assistance
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): The Intervention Group will receive 9 physical rehabilitation sessions using the MAK device. Each session will consist of approximately 90 minutes.
  Interventions: Device: Physical Rehabilitation with MAK exoskeleton

INTERVENTIONS:
Device: Physical Rehabilitation with MAK exoskeleton — The participants will assist to 9 physical rehabilitation sessions with the MAK exoskeleton. During these sessions, different movements and therapies will be conducted using the studied device.

SUMMARY:
This study aims to evaluate the safety and usability of a motorized mobility assistance exoskeleton (MAK). The procedure explores the use of the MAK exoskeleton during the static and dynamic rehabilitation sessions with the intention to evaluate the safety and usability of the device in the studied population. The protocol has been focused on defining how the device can be used appropriately in this population in a safe manner by rehabilitation specialists.The study also aims to assess the safety of clinicians implementing the intervention, as well as possible benefits derived from the use of the device. As a secondary outcome, efficacy measurements will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Weight < 100 kg
* Height between 1.5 and 1.9 meters
* Anthropometric measurements to fit in the exoskeleton:
* Distance from the center of the knee joint to the ground: 42 - 55 cm
* Distance from the center of the knee to the groin fold: more than 28 cm.
* Perimeter in thigh (midpoint trochanter - epicondyle): 40 - 63 cm.
* Perimeter in calf (point of greater volume): 30 - 44 cm.
* Ability to follow simple commands and communicate basic needs
* Presence of unilateral hemiparesis
* Diagnosis of stroke confirmed with imaging tests.
* Sub-acute or chronic patients (time since diagnosis 1 month or more)
* Score on FAC scale from 1 to 4
* Sufficient postural control to maintain standing posture and to take a step with the weight on the affected lower limb, manual assistance or technical aids being allowed

Exclusion Criteria:

* Spasticity > 3 in lower limbs according to the MAS scale
* Skin alterations in the contact areas with the exoskeleton
* Planned surgical intervention during the duration of the study
* Two or more osteoporotic fractures in the lower limbs in the last 2 years
* Presence of other pathologies that cause exercise intolerance (such as uncontrolled hypertension, coronary artery disease, arrhythmia, congestive heart failure, Parkinson's, severe lung disease)
* Surgical operation in the 3 months prior to the start of the study on the lower limbs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Safety as number of serious device adverse events | after each use of exoskeleton, for 5 weeks
  Presence of a serious device adverse events where the participant or therapist is involved

SECONDARY OUTCOMES:
Safety as presence of adverse events or adverse device events | after each use of exoskeleton, for 5 weeks
  Presence of a device adverse events where the participant or therapist is involved
Exercises [measured as time per exercise in seconds] | after each use of exoskeleton, for 5 weeks
  Measured as time per event at each therapy session
Transfers [measured as time to carry out the transfers in seconds] | At each use of exoskeleton, for 5 weeks
  Measured as time and level of assistance to carry out the transfers
Acceptability [number of participants which discontinue the participation during the trial in relation with the included participants] | at the end of the 5th week
  Measured as abandon ratio
Accessibility [number of potential participants in relation with the included participants] | at the end of the 5th week
  Measured as relation between number of participants and number of potential participants which weren't recruited
Fall Prevalence [number of falls during the using of the device] | During the use of the device, for 5 weeks
  Number of falling events ocurred from the participant or therapist
Skin integrity [number of skin injuries related to the device] | before and after each use of exoskeleton, for 5 weeks
  skin integrity measured as the number of skin injuries
Pain [VAS scale] | Before and after the use of the device, during 5 weeks
  Pain registered before and after the use of the device, by the participant and therapist
Fatigue [Borg Scale] | Before and after the use of the device, during 5 weeks
  Fatigue registered before and after the use of the device, by the participant and therapist
Spasticity [Modified Ashworth Scale] | Before and after the use of the device, during 5 weeks
  Spasticity registered before and after the use of the device
Heart rate [measured with sphygmomanometer] | Before and after the use of the device, during 5 weeks
  Number of heart beats per minute
Physical evaluation [number of physical injuries detected] | Before and after the use of the device, during 5 weeks
  Physical Evaluation as presence of tissue damage
Muscle Strength [measured with Hand Held Dynamometer in N] | At the first day, 3rd week and 5th week
  Muscle Strength measured at hip, knee and ankle muscles
ROM [measured with goniometer] | At the first day, 3rd week and 5th week
  Range of Movement
Functional Mobility [Functional Ambulation Category scale] | At the first day, 3rd week and 5th week
  Functional Mobility with and without the device
System Usability [System Usability Scale] | At the 5th week
  Measurement of System's Usability measured by the therapist
User perception of the device [QUEST 2.0] | At the 5th week
  QUEST 2.0 will be assessed by the therapist and participant
Distance covered walking [6MWT] | At the first day, 3rd week and 5th week
  6MWT recorded using the device
Device malfunction [as number and type of device malfunction] | During the use of the device, for 5 weeks
  Any device malfunction will be recorded
Particpant's stability [TUG] | At the first day, 3rd week and 5th week
  Timed Up and Go Scale
Breath Rate [Breathings per minute] | Before and after the use of the device, during 5 weeks
  Number of breaths per 1 minute
SP/DP [sphygmomanometer] | Before and after the use of the device, during 5 weeks
  Systolic and Diastolic Pressure measured in mmHg
SpO2 [pulse oximeter] | Before and after the use of the device, during 5 weeks
  SpO2 measured in %

CONTACTS AND LOCATIONS:
Locations (1):
- MarsiCare, Madrid, Arganda Del Rey, Spain

IPD SHARING:
Plan to Share IPD: No
There's no intention to share the individual participant data with researchers outside the scope of the present study. The participant data will be collected anonymized using a code for each participant. The data will be collected and stored according to the EU regulations and local laws and guidelines.